CLINICAL TRIAL: NCT01175252
Title: Time Trend Analysis of Diarrhea-related Hospitalizations and Deaths in Children < 5 Years of Age in Brazil, 1990-2010
Brief Title: Trends Over Time (1990-2010) of Diarrhoea-related Hospitalizations and Deaths in Children < 5 Years of Age in Brazil
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112368
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Diarrhoea; Gastroenteritis
Keywords: Gastroenteritis
MeSH Terms: conditions — Diarrhea; Gastroenteritis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Gastroenteritis Cohort: All children suffering with gastroenteritis
  Interventions: Other: Database analysis

INTERVENTIONS:
Other: Database analysis — Review and collect data from database

SUMMARY:
This study aims at collecting data to obtain baseline incidence and monitor trends over time in hospitalizations and deaths from all cause gastroenteritis in children <5 years of age, before and after implementation of Rotarix™ universal mass vaccination in Brazil.

DETAILED DESCRIPTION:
In this study baseline gastroenteritis related hospital discharges and mortality data from the Ministry of Health databases (DATASUS) will be compared to the current data after introduction of Rotarix™.

ELIGIBILITY:
Inclusion Criteria:

* Gastroenteritis associated hospital discharges and gastroenteritis related deaths occurring in children <5 years of age during the period analyzed and registered in the DATASUS databases will be collected for the study

Exclusion Criteria:

* Not applicable

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children <5 years of age being hospitalized due to gastroenteritis between 1998 and 2010 and deceased due to gastroenteritis between 1990 and 2009 in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of all cause gastroenteritis related hospital discharges and deaths | In post vaccine introduction period compared to pre-vaccination period (gastroenteritis related hospital discharges from 1998 to 2010, gastroenteritis related deaths from 1990 to 2009)

SECONDARY OUTCOMES:
Occurrence of all cause gastroenteritis related hospital discharges and hospital deaths by year, region and age groups | From 1998 to 2010
Occurrence of all cause gastroenteritis related deaths by year, region and age groups | From 1990 to 2009

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Belém, Pará, Brazil

REFERENCES:
- [Background] Lanzieri TM et al. The impact of rotavirus vaccination on gastroenteritis hospitalizations among children <5 years in Brazil. Abstract presented at the 6th World Congress of World Society for Pediatric Infectious Diseases (WSPID). Buenos Aires, Argentina, 18-22 November 2009.
- [Background] Lanzieri TM, Costa I, Shafi FA, Cunha MH, Ortega-Barria E, Linhares AC, Colindres RE. Trends in hospitalizations from all-cause gastroenteritis in children younger than 5 years of age in Brazil before and after human rotavirus vaccine introduction, 1998-2007. Pediatr Infect Dis J. 2010 Jul;29(7):673-5. doi: 10.1097/INF.0b013e3181da8f23. PMID 20300045
- [Background] Lanzieri TM et al. Impact of rotavirus vaccination on childhood diarrheal deaths in Brazil. Abstract presented at the 9th International Rotavirus Symposium (IRS). Johannesburg, South Africa, 2-3 August 2010.